CLINICAL TRIAL: NCT06136416
Title: Pilot Study for the Development of an Activity and Quality of Life Questionnaire for the Follow-up of Patients With Non-dystrophic Myotonia
Acronym: MNDActivLife
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-PP-15
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Non-Dystrophic Myotonia
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Non-dystrophic myotonias (Experimental)
  Interventions: Other: Questionnaire for Non-dystrophic myotonias

INTERVENTIONS:
Other: Questionnaire for Non-dystrophic myotonias — Patients will have to complete the questionnaire created specifically for their pathology, as well as an evaluation grid of the same questionnaire to assess its relevance and good understanding

SUMMARY:
Non-dystrophic myotonias (MND) are rare neuromuscular diseases caused by mutations in the voltage-dependent channels of skeletal muscles, resulting in delayed muscle relaxation after voluntary contraction. They include various conditions such as congenital myotonia, congenital paramyotonia and sodium channel myotonia. The main characteristic is myotonia, muscle stiffness accompanied by pain, fatigue and weakness. Symptoms vary in intensity, and fluctuation complicates clinical assessment.

Until now, no validated scale to assess the severity of myotonia is the subject of a consensus among neurologists. It therefore seems necessary to establish a scale to simply and quickly assess the severity of myotonia to fill this need.

The areas of this future scale were identified by the study coordinator based on existing questionnaires and scales. These areas have been validated by a scientific committee composed of expert neurologists.

The main objective of the study is to validate the adequacy and formulation of the scale questions by involving 10 patients who will complete the questionnaire twice to assess its fidelity. At the end of the study, the committee will exclude inappropriate questions. The goal is to create a reliable scale to assess the severity of myotonia.

ELIGIBILITY:
Inclusion criteria:

* Male or female, over 18 years of age;
* With genetically diagnosed non-dystrophic myotonia;
* Affiliated with a Social Security system;
* Able to read, understand and speak French
* Having expressed his non-opposition

Exclusion criteria:

* Subject participating in an interventional study with experimental drug or in the exclusion period of an interventional study;
* Pregnant or lactating women for women of childbearing age;
* Patient protected by law under guardianship or curators, or who cannot participate in a clinical study under Article L. 1121-16 of the French Public Health Code

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Evaluate the relevance of the MNDActiveLive questionnaire | The day of inclusion
  The relevance of the MNDActiveLive questionnaire will be measured using patient responses to the relevance and formulation assessment grid. Indeed, it is about evaluating the percentage of relevant questions (that is, relatively relevant, perfectly relevant and relevant). The question will be considered relevant if the percentage is higher than 80%.

SECONDARY OUTCOMES:
Evaluate the formulation of the MNDActiveLive questionnaire | The day of inclusion
  The formulation of the MNDActiveLife questionnaire will be evaluated using the percentage of well-formulated questions (i.e., satisfactorily formulated, well-formulated, perfectly formulated) and the percentage of poorly-formulated questions (i.e. poorly worded or unclear, slightly ambiguous or confusing). The question will be considered well formulated if the percentage is greater than 80%.
Identify questions to be excluded | The day of inclusion
  Questions to be excluded will be identified using the percentage of questions poorly formulated and irrelevant (poorly formulated or unclear, slightly ambiguous or may be confusing/not at all relevant, not relevant). The question will be excluded if the percentage of poorly formulated and irrelevant questions is greater than 80%.
Identify questions to rephrase | The day of inclusion
  Questions to be reformulated will be identified using the percentage of questions that are poorly formulated and relevant (i.e., poorly formulated or unclear, slightly ambiguous or that may be confusing/relatively relevant, perfectly relevant and relevant). The question will be reformulated if the percentage is greater than 80%
Assess reproducible issues | The day of inclusion and 7 days after
  The reproducibility of each question will be assessed by the percentage of patients with change in response between the response provided at inclusion and that provided 7 days later
Select questions to keep | The day of inclusion and 7 days after
  Questions to be retained will be identified using the percentage of questions that are reproducible, well formulated and relevant

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, Alpes Maritimes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amara A, Cavalli M, Ezaru A, Puma A, Garcia J, Meiran S, Parrotta A, Vicart S, Pereon Y, Salort-Campana E, Moussy M, Nadaj-Pakleza A, Villar-Quiles RN, Sacconi S. Active-NDM: Development of a patient-reported outcome questionnaire to measure the impact of non-dystrophic myotonia on activity of daily living. J Neuromuscul Dis. 2026 Feb 2:22143602251412470. doi: 10.1177/22143602251412470. Online ahead of print. PMID 41627073